CLINICAL TRIAL: NCT04481711
Title: Investigation of the Effect of Total Knee Arthroplasty on Proinflammatory Cytokine Level, Pain Severity, Functional Status, Joint Position Sense and Radiographic Findings
Brief Title: Total Knee Arthroplasty and Clinical Findings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Murat EMİRZEOĞLU, Karadeniz Technical University, Karadeniz Technical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-91
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Orthopedic Disorder; Arthropathy of Knee; Pain, Joint; Proprioception; Radiography
MeSH Terms: conditions — Musculoskeletal Diseases; Arthralgia | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Twenty-nine patients (female/male: 24/5) with grade 4 osteoarthritis were included in the study group. These patients underwent total knee arthroplasty
  Interventions: Procedure: Total Knee Arthroplasty
- Control group (No Intervention): Twenty-two patients (female/male:13/9) with <grade 4 osteoarthritis were included in the control group.

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Osteoarthritis (OA) is one of the most common chronic peripheral joint diseases increasing among the aging population.Pathogenesis is not fully known.One of the most common risk factors and causes are loss of pain and function. Knee joint osteoarthritis adversly affects the person's life quality. Total Knee Arthroplasty (TKA) is a surgical approach to restore tibiofemoral joint alignment, especially in the severe level of knee OA.
  Arms: Study group

SUMMARY:
Knee osteoarthritis is a common disease that causes pain and loss of function. Total Knee Arthroplasty (TKA) is a frequently used surgical method in the treatment of severe knee osteoarthritis. The aim of this study was to investigate the effect of TKA on IL-6, TNF-α and IL-1β cytokine levels, pain intensity at rest and walking, knee joint valgity angle,malaligment, functional status and knee joint position sense.

DETAILED DESCRIPTION:
Twenty-nine patients (female/male: 24/5) with grade 4 osteoarthritis were included in the TKA group (study group) and 22 patients (female/male:13/9) with <grade 4 osteoarthritis were included in the control group. Systemic venous blood samples of the patients were taken to evaluate the cytokine level (IL-6, TNF-α, IL-1). The Visual Analogue Scale was used to assess pain intensity, and the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) score was used to evaluate the functional status. Valgity and malaligment measurements were calculated using antero-posterior X ray Digital goniometer was used to evaluate the knee joint position sense (at 35, 55 and 70 degrees knee flexion angles). Measurements were taken once from patients in the control group, and twice in pre-op and post-op sixth weeks from study group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade 4 degeneration levels who had surgical indications between the ages of 45-75 were placed in the study group.
* Patients without surgical indication, lower than 4 OA severity included in the control group

Exclusion Criteria:

* Patients with surgical history of the ipsilateral side, neuropathic pain, loss of sensation, systemic, chronic and infectious disease were excluded from the study

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Proinflammatory cytokine level | 30 minutes
  Systemic venous blood samples were taken. IL-6, TNF-α and IL-1β cytokine levels were examined.
Pain severity | 15 minutes
  The pain intensity were evaluated by the Visuel Analog Scale.
Functional status | 30 minutes
  The Western Ontario and McMaster Universities Arthritis Index was used for functional status.
Joint position sense | 30 minutes
  Electro-goniometer was used for proprioception evaluation
Valgity angle and amount of malaligment | 30 minutes
  In this evaluation, the valgity angle and the malalingement amount were calculated on the knee antero-posterior direct X-ray imageby an experienced orthopedist

CONTACTS AND LOCATIONS:
Overall Officials: Murat Emirzeoğlu, Study Chair — Karadeniz Technical University; Arzu Erden, Study Director — Karadeniz Technical University; Kübra Canlı, Study Chair — Hacettepe University; Serap Özer Yaman, Study Chair — Karadeniz Technical University; İbrahim Pekşen, Study Chair — Karadeniz Technical University; Osman Aynacı, Study Chair — Karadeniz Technical University; Süleyman Caner Karahan, Study Chair — Karadeniz Technical University
Locations (1):
- Karadeniz Technical Üniversitesi, Trabzon, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided